CLINICAL TRIAL: NCT01576458
Title: Randomised Placebo-controlled Study of Ursodeoxycholic Acid in the Treatment of Intrahepatic Cholestasis of Pregnancy
Brief Title: Ursodeoxycholic Acid in the Treatment of Intrahepatic Cholestasis of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Titta Joutsiniemi, MD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73/180/2011; 73/180/2011 (Registry Identifier: URSODEOXYCHOLIC ACID AND INTRAHEPATIC CHOLESTASIS OF PREGNANCY)
Record Dates: First submitted 2012-02-18; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Intrahepatic Cholestasis; Pregnancy
Keywords: ursodeoxycholic acid; intrahepatic cholestasis; pregnancy
MeSH Terms: conditions — Cholestasis, Intrahepatic | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ursodeoxycholic acid (Active Comparator): 10 pregant women with intrahepatic cholestasis of pregnancy
  Interventions: Drug: ursodeoxycholic acid
- placebo (Active Comparator): 10 pregnant women with intrahepatic cholestasis of pregnancy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ursodeoxycholic acid — 450 mg/day for 14 days
  Arms: ursodeoxycholic acid
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to examine the efficacy and safety of ursodeoxycholic acid (UDCA) in the treatment of patients with intrahepatic cholestasis of pregnancy (ICP).

In the randomised (double-blind, placebo-controlled) study 20 pregnant women with ICP received (random allocation of) either 450 mg/day UDCA or placebo for 14 days during the third trimester of pregnancy. The severity of pruritus was registered. Itching scores and serum levels of alanine aminotransferase, total bile acids, estradiol, progesterone, prolactin, cholesterol, HDL-cholesterol, triglycerides, activated partial thromboplastin time (APTT), fibrinogen D-dimers (FIDD) and platelet count were assessed before the treatment and weekly thereafter. Data on pregnancy and delivery outcome was recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with intrahepatic cholestasis of pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1998-01; Primary Completion 1998-12 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
pruritus | an average of 5 weeks
  visual analogy scale (VAS): 0-10
laboratory values | an average 5 weeks
  Serum levels of alanine aminotransferases and total bile acids were assessed before the treatment and once a week thereafter at least three times or until delivery. Simultaneously serum levels of estradiol, progesterone, prolactin, cholesterol, HDL-cholesterol and triglyserides were assessed. Platelet count activated partial thromboplastin time and fibrinogen D-dimers were measured as well.

SECONDARY OUTCOMES:
Obstetrical surveillance | 2-12 weeks
  Data on pregnancy and delivery outcome was recorded and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Timonen, PhD, Study Chair — Turku University Hospital; Ulla Ekblad, PhD, Study Director — Turku University Hospital; Riitta Leino, MD, Principal Investigator — Turku University Hospital; Pertti Palo, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Joutsiniemi T, Timonen S, Leino R, Palo P, Ekblad U. Ursodeoxycholic acid in the treatment of intrahepatic cholestasis of pregnancy: a randomized controlled trial. Arch Gynecol Obstet. 2014 Mar;289(3):541-7. doi: 10.1007/s00404-013-2995-5. Epub 2013 Aug 27. PMID 23978872